CLINICAL TRIAL: NCT01704586
Title: Clinical Evaluation of a I-124 PET/CT Based Remnant Radioiodine Ablation Decision Concept in Differentiated Thyroid Cancer Using PROBE Design
Brief Title: I-124 PET/CT Based Remnant Radioiodine Ablation Decision Concept in Differentiated Thyroid Cancer
Acronym: CLERAD-PROBE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Wuerzburg (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Principal Investigator, Manuel Weber, Dr. med.., Acad. Dir., University of Wuerzburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UKW-NUK-I-124
Record Dates: First submitted 2012-10-04; First posted 2012-10-11 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-04

CONDITIONS: Differentiated Thyroid Carcinoma
Keywords: Differentiated thyroid carcinoma; PET/CT; Radioiodine Remnant Ablation; I-124; Quality of life
MeSH Terms: interventions — Iodine-124

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radioiodine (Active Comparator): Standard procedures using only I-131. All patients in this arm will have assigned I-131 ablation, followed by periodic I-131 diagnostic re-evaluations after 4-6 months as needed.
  Interventions: Radiation: Radioiodine I-131
- I-124 (Active Comparator): I-124 PET/CT guided concept following ATA guideline recommendations after total thyroidectomy. Uptake outside of thyroid bed constitutes I-131 therapy for remnant ablation and metastasis therapy based on I-124 dosimetry. Remnant mass and/or metastasis mass will be estimated by a diagnostic CT scan simultaneously while doing PET at the optimum time point 2-3 days after administration of I-124. If there is no uptake outside of thyroid bed, no ablation will follow in stage I disease according to AJCC with the possibility of lymph node involvement but no distant metastasis and no microscopical residual disease (Patient age <45y: any T, any N, M0; Patient age 45y or older: T1, N0, M0). Periodic follow-up may include I-124 PET/CT when indicated to determine whether or not another I-131 therapy has to follow. Thyroglobuline increase also constitutes I-124 PET/CT imaging.
  Interventions: Radiation: I-124

INTERVENTIONS:
Radiation: Radioiodine I-131 — Radioiodine will be used for ablation therapy, dosimetry and posttherapeutic whole body scan, as well as low dose I-131 imaging.
  Arms: Radioiodine
Radiation: I-124 — I-124 will be used for imaging to assess uptake inside and outside of thyroid bed, using PET/CT whole body scanning, followed by I-131 therapy as necessary as per protocol.
  Arms: I-124

SUMMARY:
Thyroid nodules are a common clinical problem. Epidemiologic studies have shown the prevalence of palpable thyroid nodules to be approximately 5% in women and 1% in men living in iodine-sufficient parts of the world and up to 30% in iodine deficient regions, such as Germany. The clinical importance of thyroid nodules rests with the need to exclude thyroid cancer which occurs in 5-15%. Differentiated thyroid cancer (DTC), which includes papillary and follicular cancer, comprises the vast majority (90%) of all thyroid cancers. In Germany, approximately 7,000 new cases will be diagnosed in 2011. The yearly incidence has increased from 3.6 per 100,000 in 1973 to 8.7 per 100,000 in 2002, and this trend appears to be continuing. Recurrence-free survival is generally excellent and depends on the risk group.

The role of postoperative remnant radioiodine ablation (RRIA) as the most serious question regarding the initial management of DTC still needs to be resolved even after decades of radioiodine use. American Thyroid Association directions for future research addressing these questions include:

* Better understanding of the long-term risks of radioiodine use;
* Improved risk stratification;

Randomized controlled trials are still missing in which RRIA has proven its worth as a safe and very effective treatment that results in an improved life expectancy and a reduced recurrence rate. Many observational studies lack sufficiently high evidence. Evidence grade is rated mainly on "expert level", based on non-randomized retrospective observation studies. Although RRIA in Europe is established as adjuvant standard treatment for all patients with DTC, except those with stage T1a, it remains to be shown throughout if it is beneficial for low risk and medium risk patients without metastases (M0), also known as stage I patients according to UICC/AJCC classification, accounting for 40-90% of all patients.

Blood doses due to cumulative radioiodine therapy may well exceed 2 Gy, and RRIA induces an average blood dose of 0.28 Gy to the entire body. Risks as estimated from that dose are not insignificant. The question is whether or not the condition after remnant ablation justifies such an increased risk of a secondary malignancy. The probability of causation for a pharyngeal or breast tumour can well exceed the margin of a 50% after being exposed to RRIA or consecutive I-131 diagnostic imaging to explore measureable Tg levels. Even though radioiodine therapy can benefit some patients with advanced thyroid carcinoma, it is still unknown whether the risks of RRIA outweigh any discernable benefit. Undoubtedly, quality of life may be affected by adjuvant use of I-131.

Study Hypothesis:

The I-124 study arm may have considerable benefits for the patient included in the study. These include

* enhanced tumour and risk stratification,
* avoidance of unnecessary I-131 exposure in 30-89 percent of patients who were classified with "low risk" tumour (MACIS or AMES scoring) or "stage I disease" (UICC-AJCC TNM staging system), and,
* improved quality of life at the same or better morbidity and mortality rates in the I-124 arm.

Environmental and hospital staff related benefits include prevention or saving of I-131 exposure.

This study is designed to compare effectiveness of treatments following and evaluating guideline recommendations in two assignment arms.

ELIGIBILITY:
Inclusion Criteria common for all study subjects prior to randomisation:

* Histologically confirmed new diagnosis of DTC (including Hürthle-cell carcinoma)
* Age 18-80 years
* Performance Status of 0-2
* Tumor stage T1b to T4 with the possibility of lymph node involvement and distant metastasis according to the [TNM] staging system
* One- or two stage thyroidectomy, with or without central lymph node dissection
* Patient´s written informed consent
* Ability to comply with the protocol procedures

Exclusion criteria for all study subjects prior to randomisation:

* Anaplastic or medullary carcinoma
* History of prior malignancy within the past 5 years with limited life-time expectancy, except for cured non-melanoma skin cancer, cured in situ cervical carcinoma, or other treated malignancies with no evidence of disease for at least three years.
* Positive pregnancy test or breast feeding
* Any other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation, or which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Recent iodine contamination

After Randomisation

I-124 arm:

A: Inclusion criteria for no remnant ablation (low risk DTC):

* Stage I (according to AJCC, ref. 1,33) papillary or follicular carcinoma with the possibility of lymph node involvement but no distant metastasis and no microscopical residual disease (Patient age <45y: any T, any N, M0; Patient age 45y or older: T1, N0, M0)
* I-124 uptake only in thyroid bed
* Absence of aggressive malignant histologic subtypes, including tall-cell, insular, poorly differentiated and diffuse sclerosing thyroid cancer

B: Inclusion criteria for remnant ablation (high risk DTC):

* All other [TNM] stages (stage II to stage IV C)
* Presence of aggressive malignant histologic subtypes, including tall-cell, insular, poorly differentiated and diffuse sclerosing thyroid cancer
* I-124 uptake in and outside thyroid bed

Standard arm:

-Standard I-131 ablation concept as defined for all T1b to T4 subjects.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2015-05; Primary Completion 2021-05 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Mean blood dose after complete remission | 18 months after thyroid surgery
  Both study arms result in different I-131 activity assigned to be administered, depending on remnant ablation and/or metastasis treatment decision. I-131 activity will be standard or less in the standard arm, none in the I-124 arm in patients identified as per protocol not to be administered an ablation activity.

SECONDARY OUTCOMES:
Quality of life comparison | At diagnostic re-evaluations every 4-6 months until 18 months after thyroid surgery
  Quality of life will be assessed at each visit a patient is scheduled for re-valuation, using a standardized (SF-36) questionnaire specifically adapted for differentiated thyroid carcinoma.
Comparison of morbidity and mortality (effectiveness) between the I-124 guided and the standard arm. | At diagnostic re-evaluations every 4-6 months until 18 months after thyroid surgery
  Proportion of patients within the group under I-124 PET/CT guided concept which do not need a RRIA: Because all patients subjected to standard EANM guideline procedures will firstly have RRIA, the proportion of patients can be estimated which is not subjected to unnecessary ablation by applying the I-124 PET/CT guided concept. Thus, we can estimate the proportion of patients in the experimental arm without recurrent tumour or progression (key secondary outcome).
Prognostic value of thyroglobuline | At diagnostic re-evaluations every 4-6 months until 18 months after thyroid surgery
  The prognostic value of thyroglobuline concentration will be evaluated for both study arms in correlation with tumour stage and imaging modalities.

CONTACTS AND LOCATIONS:
Overall Officials: Peter F Schneider, MD, Prof., Study Chair — University Clinic Würzburg, Department of Nuclear Medicine; Ina Binse, MD, PhD, Principal Investigator — Universiity Clinic Essen, Department of Nuclear Medicine
Locations (2):
- Germany (2):
  - Clinic of Nuclear Medicine, University Clinic Essen, Essen
  - University Clinic Würzburg, Würzburg

REFERENCES:
- [Background] American Thyroid Association (ATA) Guidelines Taskforce on Thyroid Nodules and Differentiated Thyroid Cancer; Cooper DS, Doherty GM, Haugen BR, Kloos RT, Lee SL, Mandel SJ, Mazzaferri EL, McIver B, Pacini F, Schlumberger M, Sherman SI, Steward DL, Tuttle RM. Revised American Thyroid Association management guidelines for patients with thyroid nodules and differentiated thyroid cancer. Thyroid. 2009 Nov;19(11):1167-214. doi: 10.1089/thy.2009.0110. PMID 19860577
- [Background] Luster M, Clarke SE, Dietlein M, Lassmann M, Lind P, Oyen WJ, Tennvall J, Bombardieri E; European Association of Nuclear Medicine (EANM). Guidelines for radioiodine therapy of differentiated thyroid cancer. Eur J Nucl Med Mol Imaging. 2008 Oct;35(10):1941-59. doi: 10.1007/s00259-008-0883-1. PMID 18670773
- [Background] Hay ID. Selective use of radioactive iodine in the postoperative management of patients with papillary and follicular thyroid carcinoma. J Surg Oncol. 2006 Dec 15;94(8):692-700. doi: 10.1002/jso.20696. PMID 17131429
- [Background] Hanscheid H, Lassmann M, Luster M, Thomas SR, Pacini F, Ceccarelli C, Ladenson PW, Wahl RL, Schlumberger M, Ricard M, Driedger A, Kloos RT, Sherman SI, Haugen BR, Carriere V, Corone C, Reiners C. Iodine biokinetics and dosimetry in radioiodine therapy of thyroid cancer: procedures and results of a prospective international controlled study of ablation after rhTSH or hormone withdrawal. J Nucl Med. 2006 Apr;47(4):648-54. PMID 16595499
- [Background] Tagay S, Herpertz S, Langkafel M, Erim Y, Bockisch A, Senf W, Gorges R. Health-related Quality of Life, depression and anxiety in thyroid cancer patients. Qual Life Res. 2006 May;15(4):695-703. doi: 10.1007/s11136-005-3689-7. PMID 16688502
- [Background] Lassmann M, Reiners C, Luster M. Dosimetry and thyroid cancer: the individual dosage of radioiodine. Endocr Relat Cancer. 2010 Jun 3;17(3):R161-72. doi: 10.1677/ERC-10-0071. Print 2010 Sep. PMID 20448022
- [Background] Verburg FA, Lassmann M, Mader U, Luster M, Reiners C, Hanscheid H. The absorbed dose to the blood is a better predictor of ablation success than the administered 131I activity in thyroid cancer patients. Eur J Nucl Med Mol Imaging. 2011 Apr;38(4):673-80. doi: 10.1007/s00259-010-1689-5. Epub 2011 Jan 6. PMID 21210115
- [Background] Passler C, Prager G, Scheuba C, Kaserer K, Zettinig G, Niederle B. Application of staging systems for differentiated thyroid carcinoma in an endemic goiter region with iodine substitution. Ann Surg. 2003 Feb;237(2):227-34. doi: 10.1097/01.SLA.0000048449.69472.81. PMID 12560781